CLINICAL TRIAL: NCT00126126
Title: Evidence Based Amputee Rehabilitation (EBAR) Program
Acronym: EBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A3381-R; 3019.01 (Registry Identifier: Miami VA IRB)
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Amputation Stumps; Diabetes Mellitus
Keywords: Artificial Limbs; Evidence based medicine; Exercise; Outcomes research; Physical therapy
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBAR Program (Experimental): Evidence Based Amputee Rehabilitation Program (rehabilitation program based on performance of the Amputee Mobility Predictor
  Interventions: Other: EBAR Program
- Wait List Control (No Intervention): Wait List Control Group

INTERVENTIONS:
Other: EBAR Program — Evidence Based Amputee Rehabilitation Program
  Arms: EBAR Program

SUMMARY:
The purpose of this study is to determine if an evidence based exercise intervention improves the functional mobility of diabetic amputees (single lower leg amputation) who have already completed standard rehabilitation and prosthetic training.

DETAILED DESCRIPTION:
Subjects who pass all eligibility requirements will then undergo baseline testing by an examiner who will remain blinded to subject group assignment. Baseline testing will include the AAS, six-minute walk test, and both the AMPPro and AMPnoPro.

After baseline testing has been completed, subjects will be randomly assigned to either the intervention or wait list control. Randomization will occur in blocks of 20 such that for each panel of 20 subjects, 50% will be randomized to the intervention and 50% will be randomized to wait list control. Randomization will be performed using a random-number table to assign treatment group to status to each subject's unique identification number. Randomization status will be concealed by recording status on a card that is folded in half so that the group assignment is inside the fold. The cards will be placed in envelopes bearing identification numbers. When a subject has completed all baseline measures, the envelope with that subject's ID number will be opened and the subject will be assigned to a group.

Subjects assigned to the intervention group will undergo clinical strength testing. An individualized program will be developed for each subject based on his or her AMP test results and clinical strength testing. Subjects will then attend rehabilitation sessions 3 times per week for 8 weeks. Each session will last approximately 45 minutes including any required rest periods. Subjects will perform endurance, balance and strengthening exercises at each session. Every 6th session, subjects in the intervention group will perform a six-minute walk test, AMPPro and complete the AAS questionnaire. The results of each AMPPro test will be reviewed and the therapeutic exercise program revised according.

After follow-up testing, subjects assigned to the wait list condition will be eligible to attend the 8-week rehabilitation program. Wait list subjects in the exercise phase will also receive the same exercise intervention described above. They will also perform a six-minute walk test, AMPPro and complete the AAS questionnaire every 6th session.

ELIGIBILITY:
Inclusion Criteria:

* People with unilateral transtibial amputations (TTA)
* At the lowest level of function candidates will have the ability or potential to use a prosthesis for transfers or ambulation on level surfaces at a fixed cadence. Typical of the limited and unlimited household ambulator, the majority of candidates' ability or potential for ambulation with the ability to transverse low-level environmental barriers such as curbs, stairs, or uneven surfaces (the ceiling for candidacy) will be those TTAs who have the ability to vary cadence and can ambulate within the community.
* People with a diagnosis of diabetic mellitus and/or peripheral vascular disease leading to amputation
* Persons comfortably fitted with a prosthesis for a period of at least 6 months
* Candidates who have completed the "standard" course of rehabilitation and prosthetic training
* Candidates who score in the range of 10 to 36 on the Amputee Mobility Predictor which would indicate that subjects achieved the minimum required score to be fitted with a prosthesis but they did not attain a score that is considered to be at the highest level of functioning where additional therapy would not be of significant benefit.
* Able to tolerate a moderate intensity exercise program

Exclusion Criteria:

* Persons receiving renal dialysis
* Persons with severe cardiac or pulmonary disease limiting ability to exercise including angina or poorly controlled hypertension.
* Persons with neurological disorders such as Parkinson's disease or stroke that affect ability to ambulate
* Persons with severe lower extremity arthritis
* Persons with wound on non-amputated side
* Persons experiencing problems with prosthetic fit
* Persons with poor control of diabetes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gailey, PhD, PT, Principal Investigator — Miami Veterans Affairs Healthcare System
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

REFERENCES:
- [Result] Gailey RS, Roach KE, Applegate EB, Cho B, Cunniffe B, Licht S, Maguire M, Nash MS. The amputee mobility predictor: an instrument to assess determinants of the lower-limb amputee's ability to ambulate. Arch Phys Med Rehabil. 2002 May;83(5):613-27. doi: 10.1053/apmr.2002.32309. PMID 11994800
- [Result] Gailey RS, Scoville C, Gaunaurd IA, Raya MA, Linberg AA, Stoneman PD, Campbell SM, Roach KE. Construct validity of Comprehensive High-Level Activity Mobility Predictor (CHAMP) for male servicemembers with traumatic lower-limb loss. J Rehabil Res Dev. 2013;50(7):919-30. doi: 10.1682/JRRD.2012.05.0100. PMID 24301429
- [Result] Resnik L, Borgia M. Reliability of outcome measures for people with lower-limb amputations: distinguishing true change from statistical error. Phys Ther. 2011 Apr;91(4):555-65. doi: 10.2522/ptj.20100287. Epub 2011 Feb 10. PMID 21310896
- [Derived] Gailey R, Gaunaurd I, Raya M, Kirk-Sanchez N, Prieto-Sanchez LM, Roach K. Effectiveness of an Evidence-Based Amputee Rehabilitation Program: A Pilot Randomized Controlled Trial. Phys Ther. 2020 May 18;100(5):773-787. doi: 10.1093/ptj/pzaa008. PMID 31951260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three hundred twenty six Individuals with unilateral lower limb loss were screened. Twenty agreed to participate in the study and completed the consent process.
Pre-assignment Details: Twenty individuals who met inclusion criteria completed the consent process. Eighteen were randomized to either intervention (n = 9) or wait list control (n = 9).
Groups:
- Intervention: Evidence Based Amputee Rehabilitation Program
  Exercise: Evidence Based Amputee Rehabilitation Program
- Wait-List Control Group: These individuals waited 8 weeks in order to begin the intervention.
Period: Overall Study
Arm/Group | Intervention | Wait-List Control Group
Started | 9 | 9
Completed | 9 | 7
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Those subjects who were randomized to receive the Evidence Based Amputee Rehabilitation (EBAR) Program
- Wait List Control Group: Those subjects who were randomized to the wait-list control group.
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait List Control Group | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.4) | 63.0 (7.1) | 63.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Amputee Mobility Predictor
Description: The Amputee Mobility Predictor is a reliable and valid performance-based outcome measure of prosthetic mobility. The AMP is scored from 0-47, higher scores indicating greater prosthetic mobility. The AMP can help clinicians differentiate between different functional K-levels based on as defined by the Medicare Functional Classification Level (MFCL) system. Lower limb amputees functioning at the K2 level score between 27-36 on the AMP and are classified as limited community ambulators. Those at the K3 level score between 37-42 and are typical community ambulators who have the ability to traverse environmental barriers and performing activities that are beyond simple locomotion. Individuals at the K4 level score between 43-47 which is typical of prosthetic demands of an active adult or regular athlete. The minimal detectable change for the AMP is 3.4 points.
Time Frame: 8 weeks for intervention and for wait-list control
Population: Repeated Measures ANOVA
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Intervention | Wait-List Control Group
Number analyzed (Participants) | 9 | 7
Points
  Pre-Intervention | 36.4 (4.0) | 35.3 (2.4)
  Post-Intervention | 41.7 (4.0) | 35.6 (5.4)

2. Secondary Outcome: Six-minute Walk Test
Description: The six-minute walk test (6MWT) is a measure of overall functional mobility, and cardiopulmonary and musculoskeletal endurance. It assesses the distance ambulated in 6 minutes. The 6MWT has excellent reliability for lower limb amputees and can differentiate between amputee Medicare Functional Classification Levels (MFCL).Lower limb amputees functioning at the K2 level ambulate a mean distance of 200 meters. Those at the K3 level ambulate a mean distance of 300 meters. Those at the K4 level ambulate a mean distance of 400 meters. Service Members with traumatic lower limb loss ambulate a distance of 600 meters. The minimal detectable change for the 6MWT is 45 meters.
Time Frame: 8 weeks for intervention and wait list control group
Population: Repeated Measures ANOVA
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Wait-List Control Group
Number analyzed (Participants) | 9 | 7
meters
  Pre-Intervention | 313.6 (138.9) | 262.6 (132.4)
  Post-Intervention | 387.7 (130.6) | 268.8 (157.4)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Intervention | Wait-List Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

LIMITATIONS AND CAVEATS:
Recruitment was challenging. We screened over 350 veterans and non-veterans with lower limb loss and we were only able to enroll 20.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No